CLINICAL TRIAL: NCT00833391
Title: An Open-label, Randomized, Single Dose, Five-period Crossover Study to Evaluate the Relative Bioavailability of Different Formulations of GSK1838262 in Healthy Volunteers.
Brief Title: Relative Bioavailability Study for GSK1838262 (Gabapentin Enacarbil)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 110882
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2010-03

CONDITIONS: Pharmacokinetics; Healthy Volunteer
Keywords: healthy volunteer; formulations; bioavailability; pharmacokinetics

ARMS (1):
- GSK1838262 arm (Experimental): Each subject will participate in five dosing sessions separated by at least seven days. Subjects will receive a single dose of current formulation of GSK1838262 or one of the four new formulations of GSK1838262 at each dosing session in random sequence.
  Interventions: Drug: open label

INTERVENTIONS:
Drug: open label — This is an open-label, randomized, single-dose, five-period, crossover study. All subjects will receive GSK1838262.

SUMMARY:
The purpose of this study is to evaluate the relative drug concentrations achieved with different formulations of GSK1838262 in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, five-period, crossover study to evaluate the relative drug concentrations with different formulations of GSK1838262 in healthy volunteers. Four new formulations will be tested against the current formulation to identify the most promising new formulations for further development. Each subject will participate in five dosing periods and each period will be separated by at least seven days. Blood and urine samples will be collected over the 36 hour period following each dose administration to measure the drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

* healthy, male and female subjects aged between 18 and 65 years old.
* normal body weight.
* normal ECG, vital signs and lab tests.
* normal kidney function
* agree to use acceptable contraceptive methods required.
* capable of giving written informed consent.

Exclusion Criteria:

* positive blood alcohol or urine drug test.
* positive hepatitis B/C and HIV
* donation of more than 450 mL blood within the 56 days.
* sensitivity to gabapentin
* pregnant or lactating females
* smoker
* certain medical conditions including heart disease, psychiatric disease, gastrointestinal disease, kidney or liver dysfunction
* history of seizure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
gabapentin concentrations in blood | measured up to 36 hr after dosing

SECONDARY OUTCOMES:
gabapentin concentrations in urine | measured up to 36 hr after dosing
Safety and tolerability as measured by adverse events, vital signs, ECGs and clinical laboratory tests. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States